CLINICAL TRIAL: NCT03868046
Title: Prediction of Immune-related Adverse Events Induced by Anti-CTLA4 and Anti-PD1/PDL1 Drugs by Means of a Battery of Autoantibodies. a Multicenter Prospective Observational Cohort Study
Brief Title: Autoantibodies in Treatment with Immune Checkpoint Inhibitors (AUTENTIC)
Acronym: AUTENTIC
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Hospital de Basurto (Other); Hospital Donostia (Other); Complejo Hospitalario de Navarra (Other); Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Iñigo Les Bujanda, Principal Investigator, Hospital Universitario Araba
Other Study IDs: PI2018106 (EPA-SP)
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Metastatic Cancer; Solid Organ Cancer
Keywords: Immune-related Adverse Events; Immune Checkpoint Inhibitors; Biomarkers; Autoantibodies
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Therapeutics; Immune Checkpoint Inhibitors; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and white cells (buffy coat).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with ICIs.: All enrolled patients must have been diagnosed with a cancer potentially treatable with ipilimumab, nivolumab, pembrolizumab, atezolizumab or avelumab, alone or in combination, per standard protocol.
  Interventions: Drug: Treatment with immune checkpoint inhibitors.; Diagnostic Test: Blood tests.

INTERVENTIONS:
Drug: Treatment with immune checkpoint inhibitors. — Treatment with approved immune checkpoint inhibitors, namely ipilimumab, nivolumab, pembrolizumab, atezolizumab and avelumab, alone or in combination, administered per standard protocol.
Diagnostic Test: Blood tests. — Patients will undergo ordinary blood tests obtained at specific moments predefined per protocol and extraordinary blood tests at the time of the detection of an eventual irAE.

SUMMARY:
The aim of this study is to assess the effectiveness of a battery of autoantibodies to predict the occurrence of immune-related adverse events (irAEs) in patients with cancer who will be treated with immune checkpoint inhibitors (ICIs) per standard protocol.

DETAILED DESCRIPTION:
Introduction: Treatment with ICIs is leading to a remarkable improvement in the prognosis of several types of cancer. However, the expansion of these drugs in the field of oncology is also causing the emergence of a large diversity of irAEs, whose optimal prevention and management are still to be clarified. Nowadays, there is a growing need for reliable and validated biomarkers to predict the occurrence of irAEs in patients treated with ICIs.

Purpose: To assess the effectiveness of a battery of autoantibodies available in a laboratory of autoimmunity to predict the occurrence of irAEs in patients with cancer who will be treated with ICIs per standard protocol.

Methods: A multicenter prospective observational cohort study was designed to include a total of 221 patients diagnosed with cancer amenable to treatment with ICIs. During a period of 48 weeks, patients will be controlled in the oncology outpatient clinics of five university hospitals with accredited experience in the management of immunotherapy. Immune-related adverse events will be defined and categorized according to CTCAE v. 5.0. Considering a proportion of irAEs and losses to follow-up of 25% and 5% respectively, a sample size of 221 patients was calculated to estimate an expected sensitivity of the autoantibody battery of 0.90 with a 95% confidence interval not lower than 0.75. All the participants will undergo ordinary blood tests at specific moments predefined per protocol and extraordinary blood tests at the time of the detection of an eventual irAE. Both ordinary and extraordinary samples will be frozen and stored in the biobank of each participating hospital in the form of serum and buffy coat. Once the whole cohort reaches the 24th week (intermediate analysis) and the 48th week (definitive analysis), all the samples will be centralized in the same autoimmunity laboratory for the determination of the autoantibody battery. A predictive model of irAEs will be constructed with the autoantibodies together with other potential risk factors of immune-mediated toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Initiation of treatment with a single ICI or a combination of ICIs.
2. Acceptation of an informed consent.

Exclusion Criteria:

1. Life expectancy lower than 3 months from the initiation of treatment with ICIs.
2. Proven hypersensitivity or previous allergic anaphylactic reaction induced by a specific ICI.
3. Active autoimmune disease with severe involvement.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3.
5. Ongoing immunosuppressive therapy: prednisone at doses >10 mg/day or equivalent (>1.5 mg/day of dexamethasone), and/or any dose of azathioprine, methotrexate, mycophenolate, cyclophosphamide, leflunomide, rituximab, anti-tumor necrosis factor drugs (infliximab, etanercept, adalimumab, golimumab), belimumab and abatacept.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with cancer amenable to treatment with ICIs will be considered eligible. Potential candidates will be identified and consecutively included in the oncology outpatient clinics of five university hospitals in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-08-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of irAEs. | At 48 weeks from the initiation of ICIs.
  An irAE was defined as any symptom, sign, syndrome or disease attributable to an immune activation mechanism during an ongoing treatment with an ICI or a combination of ICIs, provided that an infectious cause and/or tumor progression have been ruled out.

SECONDARY OUTCOMES:
irAE-free survival. | At 24 weeks and at 48 weeks from the initiation of ICIs.
  Time in months from the initiation of therapy with ICIs until the occurrence of an irAE or until the date of the last follow-up.
Progression-free survival. | At 24 weeks and at 48 weeks from the initiation of ICIs.
  Time in months from the initiation of therapy with ICIs until the date of proven tumor progression or until the date of the last follow-up.
Overall survival. | At 24 weeks and at 48 weeks from the initiation of ICIs.
  Time in months from the initiation of therapy with ICIs until the date of patient's death or until the date of the last follow-up.
Incidence of development of autoantibodies. | At 24 weeks and at 48 weeks from the initiation of ICIs.
  Positive conversion of the autoantibody battery after the initiation of therapy with ICIs.

CONTACTS AND LOCATIONS:
Overall Officials: Iñigo Les Bujanda, MD PhD, Principal Investigator — Hospital Universitario Araba
Locations (1):
- Hospital Universitario Araba, Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be available for exploitation in future research projects. This statement also includes the availability of the study protocol, the statistical analysis plan, the informed consent form, the clinical study report and the analytic code.